CLINICAL TRIAL: NCT03145025
Title: An Observational Change-From-Baseline Evaluation of Corneal Endothelial Cell Density in Eyes Treated With a Fluocinolone Acetonide Intravitreal Implant
Brief Title: Corneal Endothelial Cell Density in Eyes Treated With a Fluocinolone Acetonide Intravitreal Implant
Status: Completed | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 853
Record Dates: First submitted 2017-04-25; First posted 2017-05-09 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Uveitis, Posterior
MeSH Terms: conditions — Uveitis, Posterior | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Retisert — Intravitreal Implant
Drug: Fluocinolone Acetonide Intravitreal Implant — Intravitreal Implant

SUMMARY:
An Observational Change-From-Baseline Evaluation of Corneal Endothelial Cell Density in Eyes Treated with a Fluocinolone Acetonide Intravitreal Implant

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, single arm, observational evaluation of the corneal ECD change from baseline for subjects having the Retisert FA drug delivery system (0.59 mg) surgically implanted in the ocular vitreous chamber of at least 1 previously unimplanted eye for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Are scheduled for surgical placement of a Retisert fluocinolone acetonide (FA) intravitreal implant in a previously unimplanted eye.
2. Are able and willing to comply with all treatment and follow up/study procedures.
3. Able and willing to provide informed consent or, for subjects 12-18 years of age, have the ability to understand and provide assent (when applicable) and whose parent/legally authorized representative has the ability to understand and provide written informed consent on the Institutional Review Board (IRB) approved informed consent form (ICF) and provide authorization as appropriate for local privacy regulations.
4. For female subjects:

Note: Should a subject conceive during the study, the pregnancy should be reported as soon as possible to the study Medical Monitor and Promedica International within 24 hours. The pregnancy will be followed up to term. The subject will continue in the studyregardless if pregnancy is reported on an AE/SAE form. If an Investigator becomes aware of a post study pregnancy 30 days after the study exit visit while Fluocinolone Acetonide Implant remains in the subject's study eye, then it should be reported as a post-marketing report

Exclusion Criteria:

1. Has previously, concurrently or anticipated enrollment in Bausch & Lomb study 440, titled, "An Observational Bilateral Evaluation of Corneal Endothelial Cell Density in Subjects Who Have Had a Fluocinolone Acetonide Implant for at Least One Year."
2. Has severe/serious ocular pathology or medical condition that could result in the subject's inability to complete the study, based on the judgment of the Investigator.
3. Has participated in an ophthalmic drug or device research study within 30 days prior to Screening (Visit 1, Day -30 to -1) in this study
4. Is monocular (unable to detect hand motion at 6 feet in 1 eye).
5. Has a known corneal dystrophy or corneal transplant.
6. Has a history of ocular surgery in the eye scheduled for implant surgery, including laser procedures, within the 30 days prior to Screening (Visit 1, Day -30 to -1).
7. Had any type of intraocular drug delivery implant (eg, Retisert, Ozurdex [dexamethasone intravitreal implant]) in the study eye.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects having the Retisert FA drug delivery system (0.59 mg) surgically implanted in the ocular vitreous chamber of at least 1 previously unimplanted eye for at least 1 year
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint is change from baseline in endothelial cell density (ECD) in the study eye one year following implantation. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Valeant Site 001, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes